CLINICAL TRIAL: NCT03145376
Title: Clinical Evaluation and Geriatric Assessment in Elderly Patients Before and After Percutaneous Aortic Valve Implantation (TAVI) or MitraClip Positioning
Brief Title: Clinical and Geriatric Assessment in Elderly Patients Before and After TAVI or MitraClip Positioning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Piccirillo, associate professor, University of Roma La Sapienza
Other Study IDs: TaMi01
Record Dates: First submitted 2017-03-27; First posted 2017-05-09 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Mitral Valve Insufficiency; Aortic Stenosis Senile
Keywords: TAVI; MitraClip; geriatric assessment; heart rate variability; elderly
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients before and after TAVI/MitraClip: geriatric assessment of patients before and after TAVI/Mitraclip
  Interventions: Diagnostic Test: geriatric assessment

INTERVENTIONS:
Diagnostic Test: geriatric assessment — 1. Clinical evaluation and geriatric assessment with:
     1. CIRS: CIRS (Cumulative Illness Rating Scale)
     2. ADL (Activities of Daily Living);
     3. IADL (InstrumentalActivities of Daily Living);
     4. Mini Nutritional Assessment;
     5. Evaluation of quality of life (Short Form 36, SF-36).
  2. Making a traditional 12-lead ECG.
  3. A single lead electrocardiographic registration (DI, D II and D III) of 5 minutes baseline and 5 minutes with controlled breathing (15 breaths / min), using the Spectralink 2011 program, which allows us to identify and calculate the variables object of study;
  4. transthoracic echocardiogram.
  Other Names: ECG; Heart Rate Variability; Echocardiogram

SUMMARY:
Since October of 2014, the Policlinico Umberto I Hospital has an "Heart Team", a group of selected specialists with the task of assessing and identifying eligible patients for valvular aortic transcatheter implantation (TAVI) or a placement of a MitraClip .

The specialists taking part to Heart Team are: a cardiologist, a heart surgeon, a vascular surgeon, an anesthesiologist and a geriatrician.

The Geriatrician is called to make a careful multidimensional assessment of the elderly patients who have been suggested for the interventions mentioned above. His role is to assess the degree of co-morbidity and polypathology, autonomy in the common activities of daily living, nutritional status, cognitive status and quality of life. Following this evaluation, together with the other components of Heart Team, it is expressed a collective judgment on the patient's eligibility to these interventions. So, the aim of the present study is to identify changes in the degree of cognitive decline, of autonomy in carrying out activities of daily living, quality of life, nutritional status, pre- and postoperatively (6 months after the procedure) polypathology degree in elderly patients to be undergone or undergoing TAVI or positioning MitraClip because suffering from aortic valvular stenosis or severe mitral insufficiency. The patients undergo to a battery of tests, to a 5 minutes electrocardiographic record to evaluate the Heart Rate Variability (HRV) and to a complete echocardiographic evaluation.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a progressive chronic valvular disease that progressively and rapidly leads to the development of heart failure. This pathology, which is typical of the elderly, is increasing together with the age of the population and it is a candidate for the development of less invasive and innovative therapies that enable the treatment of older patients with polypathology and high degree of comorbidity. According to the most recent guidelines for the treatment of valvular heart disease, the degenerative AS is the most common valve disease in Western countries especially in the group aged over 65 years. The degenerative AS, in its most severe form, is a highly debilitating chronic condition characterized by symptoms as such precordial pain suggestive of angina, transient altered state of consciousness, or syncope, dyspnea and other heart failure symptoms secondary to reduced stroke volume. A recent systematic review (2) estimated the prevalence of AS in the elderly population aged over 75 years amounted to 12.4% while the prevalence of severe AS amounted to 3.4%. The average survival after the onset of symptoms is about 2-3 years. The natural history of the disease is not modified by conservative treatment and, to date, the surgical aortic valve replacement is recommended by both the American and European guidelines for patients with severe symptomatic and asymptomatic patients with reduced ejection fraction (80 years obtain appreciable results with a less than 10% mortality and morbidity between 5 and 10%. Some conditions, such as the presence of comorbidities (chronic obstructive pulmonary disease, vasculopathy, chronic renal failure, dementia and other) and the advanced age of the patients, make the surgery too risky or impossible to achieve. Therefore, approximately one third of patients in advanced age is not currently subjected to surgery.

After the "first man" made in 2002, TAVI has been introduced in the clinic in 2007 and has quickly gained critical acclaim. Up to now, about 150,000 TAVI procedures were performed with a growing trend.

The methodical approach of the techniques involve various approaches: transfemoral, transapical, (the two most popular), transaxillary, transaortic.

The enormous diffusion of the method follows the growing demand. Conservative treatment of the SA guarantees any improvement; optimized drugs therapy is able nor to mitigate the symptomatology associated nor to resolve the underlying disease.

The surgery requires the use of extracorporeal circulation and, although conducted in the less invasive way possible, it remains an intervention in which elderly patients with polypathology and high degree of comorbidity are hardly addressed.

A clinical evaluation and multidimensional geriatric assessment are indispensable to ensure a correct diagnosis of the patient, estimating the risk of periprocedural mortality and morbidity and evaluate the actual possibility of intervention benefit on the patient's overall health.

MitraClip

The severe mitral regurgitation is a clear indication to intervention of mitral repair which has advantages compared to traditional surgery, preserving the contractile function of the left ventricle, reducing the incidence of adverse events related to the system of the prosthesis, by reducing the hospital mortality, morbidity and hospitalization, improving the long-term survival. The surgical risk of mitral plastic surgery presents a percentage lower than 2.5% in the centers that perform no less than 140 operations per year. However, an ejection fraction (FE) of the left ventricle lower than 55% is a negative prognostic index. In addition, the mitral plastic surgery has a long and difficult learning curves, but also the indisputable advantage of less invasiveness than traditional surgery, which allows its use even in patients deemed to be at higher operative risk. The placement of a MitraClip is the evolution of conventional surgery (Alfieri's speech): percutaneous, trans-septal puncture, placing clips on the mitral leaflets to create a dual orifice and therefore decrease or completely abolish the valve insufficiency . The EVEREST II study has shown that this procedure is less effective than surgery in reducing the degree of mitral regurgitation, but the percutaneous repair of mitral regurgitation is more secure and has shown improved clinical outcomes, comparable to cardiac surgery. At a post-hoc analysis, patients who benefit most from the MitraClip patients are elderly with low ejection fraction and functional mitral insufficiency. Considering that the prevalence of mitral insufficiency in the elderly is 30-50%, it is comprehensible how the MitraClip will have certain evolution in numerical terms.

The MitraClip is, therefore, a valid therapeutic option in case of functional mitral regurgitation, since the surgery in these patients is burdened with high mortality, by high recurrence of mitral regurgitation and a long hospital stay.

The MitraClip is to be used in a small number of properly selected patients. The procedural success depends on the ability to choose an individualized therapy for each patient depending on valvular anatomy, valve functionality, on comorbidities and on patient's life expectation, performing an estimation of the risk-benefit of the two percutaneous techniques and surgical intervention.

This estimate and evaluation of the patient must be operated in the geriatric multidisciplinary field, to ensure a comprehensive risk assessment of patients and their best selection.

Aim of the study

Identify changes in the degree of cognitive decline, of autonomy in carrying out activities of daily living, quality of life, nutritional status, pre- and postoperatively (6 months after the procedure) polypathology degree in elderly patients to be undergone or undergoing TAVI or positioning MitraClip because suffering from aortic valvular stenosis or severe mitral insufficiency. The patients undergo to a battery of tests, to a 5 minutes electrocardiographic record to evaluate the Heart Rate Variability (HRV) and to a complete echocardiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than or equal to 65 aa;
* the capacity to perform geriatric assessment tests;
* sinus rhythm at the time of evaluation (for the evaluation of HRV only);
* to sign appropriate informed consent.

Exclusion Criteria:

* altered cognitive abilities such as to impair the evaluation;
* hemodynamically unstable patient;
* Inability or unwillingness to sign informed consent.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients with severe aortic stenosis eligible for TAVI or affected by mitral valve severe insufficiency treatable by MitraClip positioning.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive impairment evaluation using minimental state examination (MMSE) | Baseline evaluation and a new one after 6 months to evaluate possible changes
  evaluation of the pre and post-operative cognitive impairment using the same test (mini mental state examination, MMSE: tot 28-30 points no cognitive impairment, 24-27 borderline, 19-23 mild cognitive impairment, 14-18 moderate cognitive impairment, <14 severe cognitive impairment)

SECONDARY OUTCOMES:
Quality of Life | Baseline evaluation and a new one after 6 months
  evaluation of the pre- and post-operative patient's quality of life with SF36 scale: 2 cumulative scores for physical and mental health
polypathology status evaluation with CIRS scale | Baseline evaluation and a new one after 6 months
  Cumulative Illness Rating Scale: ICS and ICC, cumulative final score can vary theoretically vary from 0 to 56
ADL: Activities of Daily Living | Baseline evaluation and a new one after 6 months
  Rating capability to attend 6 Activities of Daily Living (Have shower; Dressing; Going to the toilet; urinary incontinence; walking; having meal: tot score 0-6)
IADL:InstrumentalActivities of Daily Living | Baseline evaluation and a new one after 6 months
  rating capability to perform Instrumental Activities of Daily Living: using phone, shopping food, using means of transport, taking therapy, money management (for male and female) and doing laundry, doing housework and preparing meal evaluated just for female.
MNA:Mini Nutritional Assessment | Baseline evaluation and a new one after 6 months
  Evaluation of nutritional status with mini nutritional assessment score: max 30 points (optimal nutritional status)
mortality | phone call after 6 months from baseline evaluation
  time death after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Piccirillo, MD, PhD, Principal Investigator — Sapienza
Locations (2):
- Italy (2):
  - Gianfranco Piccirillo, Rome
  - Policlinico Umberto I, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piccirillo G, Moscucci F, Mastropietri F, Di Iorio C, Mariani MV, Fabietti M, Stricchiola GM, Parrotta I, Sardella G, Mancone M, Magri D. Possible predictive role of electrical risk score on transcatheter aortic valve replacement outcomes in older patients: preliminary data. Clin Interv Aging. 2018 Sep 11;13:1657-1667. doi: 10.2147/CIA.S170226. eCollection 2018. PMID 30237702